CLINICAL TRIAL: NCT06445062
Title: A Platform Study of RAS(ON) Inhibitors in Patients With Gastrointestinal Solid Tumors
Brief Title: Study of RAS(ON) Inhibitors in Patients With Gastrointestinal Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-GI-102
Record Dates: First submitted 2024-05-20; First posted 2024-06-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; CRC; Pancreatic Ductal Adenocarcinoma; PDAC; Gastrointestinal Cancer; Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: CRC; PDAC; RAS Mutation; KRAS G12X; Colorectal Cancer; Pancreatic Cancer; Pancreatic Ductal Carcinoma; KRAS Q61 Mutation; KRAS G12 Mutation; RAS Wild-type; RAS G12D Mutation
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal | interventions — Bevacizumab; Cetuximab; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Subprotocol A: RAS-mutated unresectable or metastatic CRC or metastatic PDAC (Experimental): RMC-6236 (QD) and Bevacizumab with 5-fluorouracil-based regimens
  Interventions: Drug: RMC-6236; Drug: mFOLFOX6 regimen; Drug: bevacizumab; Drug: mFOLFIRINOX regimen
- Subprotocol B: RAS-mutated unresectable or metastatic CRC or metastatic PDAC (Experimental): RMC-6236 (QD) and Cetuximab with or without mFOLFOX6
  Interventions: Drug: RMC-6236; Drug: mFOLFOX6 regimen; Drug: cetuximab
- Subprotocol C: metastatic PDAC (Experimental): RMC-6236 (QD) and Gemcitabine with Nab-paclitaxel
  Interventions: Drug: RMC-6236; Drug: gemcitabine; Drug: nab-paclitaxel
- Subprotocol D: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC (Experimental): RMC-9805 (QD or BID) with or without RMC-6236 (QD), and Bevacizumab with 5-fluorouracil- based regimens
  Interventions: Drug: RMC-6236; Drug: mFOLFOX6 regimen; Drug: bevacizumab; Drug: mFOLFIRINOX regimen; Drug: RMC-9805
- Subprotocol E: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC (Experimental): RMC-9805 (QD or BID) with or without RMC-6236 (QD), and Cetuximab with or without mFOLFOX6
  Interventions: Drug: RMC-6236; Drug: mFOLFOX6 regimen; Drug: cetuximab; Drug: RMC-9805
- Subprotocol F: RAS G12D-mutated metastatic PDAC (Experimental): RMC-9805 (QD or BID) with or without RMC-6236 (QD), and Gemcitabine with Nab-paclitaxel
  Interventions: Drug: RMC-6236; Drug: gemcitabine; Drug: nab-paclitaxel; Drug: RMC-9805

INTERVENTIONS:
Drug: RMC-6236 — Oral tablet
Drug: mFOLFOX6 regimen — IV infusion
  Arms: Subprotocol A: RAS-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol B: RAS-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol D: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol E: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC
Drug: bevacizumab — IV infusion
  Arms: Subprotocol A: RAS-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol D: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC
Drug: mFOLFIRINOX regimen — IV infusion
  Arms: Subprotocol A: RAS-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol D: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC
Drug: cetuximab — IV infusion
  Arms: Subprotocol B: RAS-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol E: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC
Drug: gemcitabine — IV infusion
  Arms: Subprotocol C: metastatic PDAC; Subprotocol F: RAS G12D-mutated metastatic PDAC
Drug: nab-paclitaxel — IV infusion
  Arms: Subprotocol C: metastatic PDAC; Subprotocol F: RAS G12D-mutated metastatic PDAC
Drug: RMC-9805 — Oral Tablet
  Arms: Subprotocol D: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol E: RAS G12D-mutated unresectable or metastatic CRC or metastatic PDAC; Subprotocol F: RAS G12D-mutated metastatic PDAC

SUMMARY:
The purpose of this platform study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of novel RAS(ON) inhibitors combined with Standard(s) of Care (SOC) or with novel agents.

The current subprotocols include the following:

Subprotocol A: RMC-6236 + 5-fluorouracil-based regimens

Subprotocol B: RMC-6236 + cetuximab with or without mFOLFOX6

Subprotocol C: RMC-6236 + gemcitabine + nab-paclitaxel

Subprotocol D: RMC-9805 with or without RMC-6236 + 5-fluorouracil-based regimens

Subprotocol E: RMC-9805 with or without RMC-6236 + cetuximab with or without mFOLFOX6

Subprotocol F: RMC-9805 with or without RMC-6236 + gemcitabine + nab-paclitaxel

DETAILED DESCRIPTION:
The platform study design allows combinations of RAS(ON) inhibitors with other anticancer agents to be evaluated in patients with RAS-mutated solid tumors with a focus on GI cancers.

This is an open-label platform study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of novel RAS(ON) inhibitors combined with Standard of Care (SOC) or with novel agents, and to define the Recommended Phase 2 Dose and Schedule (RP2DS). Enrollment of patients with RAS mutations will be specified in each subprotocol.

Subprotocol A is an open-label, multicenter study of RMC-6236 in combination with 5-fluorouracil-based regimens in patients with treatment-naïve unresectable or metastatic colorectal cancer or treatment-naïve metastatic pancreatic ductal adenocarcinoma. Subprotocol B is an open-label, multicenter study of RMC-6236 in combination with cetuximab with or without mFOLFOX6 in patients with unresectable or metastatic colorectal cancer or patients with previously treated or treatment-naïve metastatic pancreatic ductal adenocarcinoma. Subprotocol C is an open-label, multicenter study of RMC-6236 in combination with gemcitabine and nab-paclitaxel in patients with treatment-naïve metastatic pancreatic ductal adenocarcinoma. Subprotocol D is an open-label, multicenter study of RMC-9805 with or without RMC-6236 in combination with 5-fluorouracil-based regimens in patients with RAS G12D-mutant unresectable or metastatic colorectal cancer or metastatic pancreatic ductal adenocarcinoma. Subprotocol E is an open-label, multicenter study of RMC-9805 with or without RMC-6236 in combination with cetuximab-based therapies with or without mFOLFOX6 in patients with RAS G12D-mutant unresectable or metastatic colorectal cancer or metastatic pancreatic ductal adenocarcinoma. Subprotocol F is an open-label, multicenter study of RMC-9805 with or without RMC-6236 in combination with gemcitabine and nab-paclitaxel in patients with RAS G12D-mutant metastatic pancreatic ductal adenocarcinoma.

Each subprotocol consists of two parts: Part 1 - Dose Exploration and Part 2 - Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

All Patients (unless otherwise noted):

* ≥ 18 years of age
* ECOG PS is 0 to 1
* Adequate organ function as outlined by the study
* Pathologically or cytologically documented pancreatic carcinoma or poorly differentiated pancreatic carcinoma with metastatic disease or RAS-mutated, histologically or cytologically confirmed colorectal adenocarcinoma with documented unresectable or metastatic disease (Subprotocol A, B, and C)
* Presence of RAS G12D mutation (Subprotocol D, E, F)

Exclusion Criteria:

All Patients:

* Primary central nervous system (CNS) tumors
* Impaired gastrointestinal (GI) function that may significantly alter the absorption of RMC drugs
* Major surgery within 28 days of first dose

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1130 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 3 years
  Evaluate the safety and tolerability in the study population characterized by incidence, abnormal laboratory assessments, severity, and seriousness of adverse events in relation to the study treatment.
Dose limiting toxicities | 28 days
  Number of participants with dose limiting toxicities

SECONDARY OUTCOMES:
Pharmacokinetics of RMC-6236 and RMC-9805 | 21 weeks
  Blood concentration of RMC-6236 and RMC-9805 over time
ORR | Up to 3 years
  Overall Response Rate per RECIST v1.1
DOR | Up to 3 years
  Duration of Response per RECIST v1.1
DCR | Up to 3 years
  Incidence of Response per RECIST v1.1
TTR | Up to 3 years
  Time to Response per RECIST v1.1
PFS | Up to 3 years
  Progression Free Survival per RECIST v1.1
OS | Up to 3 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Revolution Medicines
Locations (32):
- United States (32):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Cancer at Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology- Santa Monica, Los Angeles, California
  - University of Colorado Hospital-Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale-New Haven Hospital-Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Clinical Research Center, Westwood, Kansas
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Atlantic Health System, Morristown, New Jersey
  - Northwell Health / RJ Zuckerberg Cancer Center, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center Main Campus, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Dallas, Irving, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Cregg J, Edwards AV, Chang S, Lee BJ, Knox JE, Tomlinson ACA, Marquez A, Liu Y, Freilich R, Aay N, Wang Y, Jiang L, Jiang J, Wang Z, Flagella M, Wildes D, Smith JAM, Singh M, Wang Z, Gill AL, Koltun ES. Discovery of Daraxonrasib (RMC-6236), a Potent and Orally Bioavailable RAS(ON) Multi-selective, Noncovalent Tri-complex Inhibitor for the Treatment of Patients with Multiple RAS-Addicted Cancers. J Med Chem. 2025 Mar 27;68(6):6064-6083. doi: 10.1021/acs.jmedchem.4c02314. Epub 2025 Mar 8. PMID 40056080